CLINICAL TRIAL: NCT00624234
Title: Neurobiology and Treatment of Reading Disability in Neurofibromatosis Type 1 (NF-1)
Brief Title: Neurobiology and Treatment of Reading Disability in NF-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Laura Cutting, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS049096 (NIH); NF1-R01; R01NS049096 (NIH)
Record Dates: First submitted 2008-02-25; First posted 2008-02-27 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Neurofibromatosis Type 1; Reading Disabilities
Keywords: neurofibromatosis type 1; reading disabilities; NF-1; learning disabilities; tutoring intervention
MeSH Terms: conditions — Neurofibromatosis 1; Dyslexia; Learning Disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- NF-Tutoring Program 1 (Experimental): Tutoring Program I
  Interventions: Behavioral: Tutoring Program I
- NF-Tutoring Program 2 (Experimental): Tutoring Program II
  Interventions: Behavioral: Tutoring Program II
- Typically Developing Readers (No Intervention): Control group
- IRD-Tutoring Program 1 (Experimental): Tutoring Program I
  Interventions: Behavioral: Tutoring Program I
- IRD-Tutoring Program 2 (Experimental): Tutoring Program II
  Interventions: Behavioral: Tutoring Program II
- Waitlist Control (No Intervention): Intervention Control Group (RD)

INTERVENTIONS:
Behavioral: Tutoring Program I — Tutoring Program I is a structured multi-sensory program that is designed to gradually present the range of sounds and letters with focus on accuracy of phonological concepts and application of those concepts in phrases and sentences. The instruction uses a sequenced defined lesson plan with accuracy and automaticity criteria for skill progression. A range of manipulative and kinesthetic activities is outlined to maintain learner engagement in the intensive intervention design.
  Arms: IRD-Tutoring Program 1; NF-Tutoring Program 1
Behavioral: Tutoring Program II — Tutoring Program II is designed to teach visual and speech elements of reading separately at first, and then bring them together for maximum efficiency. The program uses the idea of teaching concepts about the structure of words. For example, students transfer the rules they have learned about one vowel or structure to another without specific instructions on the new one. Tutoring Program II incorporates pictures and activities to help remember strategies for increasing basic reading skills. Speed drills are also used for development of decoding automaticity.
  Arms: IRD-Tutoring Program 2; NF-Tutoring Program 2

SUMMARY:
The goal of this trial is to determine if children with neurofibromatosis type 1 who have reading disabilities respond the same way-both behaviorally and neurobiologically-to specialized treatment programs as children with idiopathic reading disabilities do, and to determine which intervention is best for particular learner profiles.

DETAILED DESCRIPTION:
The most common concern of parents of children with neurofibromatosis type 1 (NF-1) is learning disabilities (LD). Approximately one half of all children with NF-1 have LD-the most debilitating and common of which are reading disabilities.

The purpose of this study is to determine if children with NF-1 who have reading disabilities respond the same way-both behaviorally and neurobiologically-to specialized treatment programs known to improve the decoding deficits in children with idiopathic reading disabilities. The trial will also determine which intervention is best for particular learner profiles. The overall purpose of this research is to gain a deeper understanding of the characteristics and treatment of reading disabilities in NF-1.

In the trial, researchers will compare children with NF-1 who show weaknesses in reading to children with reading disabilities of no known cause (idiopathic) using two different interventions and behavioral and neurobiological measures. Both interventions focus on teaching sound-symbol relationships, but vary in terms of relative emphasis on verbal versus visual methods of teaching.

Scientists hope findings from the trial will advance knowledge about the best therapies for LD in children with NF-1. And, by further refining how children with NF-1 who have reading disabilities are similar (or different) to children with idiopathic reading disabilities, the researchers may be able to learn if reading interventions that address areas other than decoding will also benefit children with NF-1. Also, by understanding the similarities and/or differences in the neuropsychological and neurobiological profiles of children with NF-1 who have reading disabilities, and those without, scientists will be able to refine the cognitive phenotype and neurobiological characteristics of NF-1, which will further understanding of central nervous system abnormalities in NF-1.

ELIGIBILITY:
Inclusion Criteria:

This study will be open to all individuals, ages 8 to 17 years, who meet eligibility criteria regardless of race, gender, or socioeconomic status.

* The Reading Disabilities group (including those with NF-1) is defined by scoring equal to or less than the 25th percentile on measures of basic word reading skills.
* The Control group (including those with NF1) is defined by scoring equal to or above the 40th percentile on the average of the Letter Word Identification and Word Attack subtests from the WJ-III.

Exclusion Criteria:

Any child, regardless of which group he/she is recruited for, will be excluded if he/she meets any of the following criteria (determined during phone screening, medical review, and during testing):

* is in foster care;
* previous diagnosis of mental retardation;
* known uncorrectable visual impairment;
* history of known neurological disorder (e.g., epilepsy, spina bifida, cerebral palsy, traumatic brain injury);
* documented hearing impairment greater than 25 dB loss in either ear;
* medical contraindication to MRI procedures, if participating in MRI (including exposure to metal and pregnancy);
* individuals known to have an IQ below 70;
* history or presence of a pervasive developmental disorder;
* during the DICA-IV parents indicate the presence of any severe psychiatric diagnoses or pervasive developmental disorder.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie E. Cutting, Ph.D., Principal Investigator — Vanderbilt University Special Education Department; Martha Bridge Denckla, M.D., Principal Investigator — Kennedy Krieger Institute, Johns Hopkins University, Johns Hopkins University School of Medicine; Sheryl L. Rimrodt, M.D., Principal Investigator — Vanderbilt University Pediatrics Department; John Gore, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Vanderbilt University Institute of Imaging Science, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified behavioral data (Woodcock Johnson-III NU scores) may be shared with other researchers upon request. De-identified T1 structural neuroimaging scans will be shared with other researchers through a neuroimaging data warehouse or consortium.

REFERENCES:
- See also: Additional study information — https://ebrl.vkcsites.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was 2006-2012 and was done via NF organizations and NF clinics, as well as the community recruitment.
Pre-assignment Details: Exclusions: Incomplete Data (n=31), NF without Reading Difficulty (n=11), Age (n=13; excluded CNT and RD age 15yr and over because no NF-RD over 14yr), Low IQ (n=2), Ineligible (n=12; did not fit criteria for either RD or CNT group), Prior to Intervention Change (n=26; enrolled prior to an NIH-approved change in study design regarding intervention)
Groups:
- Typically Developing Readers: Control group--children who do not have reading problems
- IRD- Tutoring Program 1: These are children with reading disabilities (without NF - ideopathic reading disabilities; IRD) who received Tutoring Program I
  Tutoring Program I: Tutoring Program I is a structured multi-sensory program that is designed to gradually present the range of sounds and letters with focus on accuracy of phonological concepts and application of those concepts in phrases and sentences. The instruction uses a sequenced defined lesson plan with accuracy and automaticity criteria for skill progression. A range of manipulative and kinesthetic activities is outlined to maintain learner engagement in the intensive intervention design.
- IRD-Tutoring Program 2: These are children with reading disabilities (without NF - ideopathic reading disabilities; IRD) who received Tutoring Program II
  Tutoring Program II: Tutoring Program II is designed to teach visual and speech elements of reading separately at first, and then bring them together for maximum efficiency. The program uses the idea of teaching concepts about the structure of words. For example, students transfer the rules they have learned about one vowel or structure to another without specific instructions on the new one. Tutoring Program II incorporates pictures and activities to help remember strategies for increasing basic reading skills. Speed drills are also used for development of decoding automaticity.
- Waitlist Control: These are children who have reading disabilities (without NF) but did not receive intervention until after the trial.
Period: Overall Study
Arm/Group | NF-Tutoring Program 1 | NF-Tutoring Program 2 | Typically Developing Readers | IRD- Tutoring Program 1 | IRD-Tutoring Program 2 | Waitlist Control
Started | 8 | 9 | 26 | 14 | 18 | 14
Completed | 8 | 9 | 26 | 14 | 18 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants both with and without NF1 were determined by researcher-administered assessments as having Reading Difficulties or typically developing reading skills.
Groups:
- Total: Total of all reporting groups
Arm/Group | NF-Tutoring Program 1 | NF-Tutoring Program 2 | Typically Developing Readers | IRD- Tutoring Program 1 | IRD-Tutoring Program 2 | Waitlist Control | Total
Number analyzed (Participants) | 8 | 9 | 26 | 14 | 18 | 14 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.62 (1.13) | 11.06 (1.48) | 9.70 (1.53) | 10.08 (1.63) | 10.33 (2.12) | 10.72 (2.25) | 10.18 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 13 | 6 | 9 | 3 | 37
  Male | 3 | 8 | 13 | 8 | 9 | 11 | 52
Woodcock Johnson Achievement Tests [Mean (Standard Deviation); unit: units on a scale] — This metric measures reading abilities (word recognition and decoding) as assessed by standard educational assessments (Woodcock Johnson Psychoeducational Battery - 3rd Edition Normative Update; WJ-III NU). The scores are reported as age-normed standard scores, with higher scores reflecting better performance on the measure (mean=100, standard deviation=15, such that a score >130 would be very superior and a score <70 would be very low). The Basic Reading score is a normed composite of the WJ-III subtests Letter-Word Identification and Word Attack, representing word-level reading skill.
  units on a scale | 78.25 (9.05) | 85.78 (7.24) | 103.81 (7.41) | 77.57 (13.47) | 79.67 (9.59) | 79.64 (9.66) | 86.88 (14.48)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WJ-III Basic Reading Normative Update (Woodcock Johnson Psychoeducational Battery - 3rd Edition; WJ-III NU) Standard Score at 15 Hours
Description: This metric measures change in reading abilities, including word recognition and decoding, as assessed by standard educational assessments (Woodcock Johnson Psychoeducational Battery - 3rd Edition Normative Update; WJ-III NU). The scores are reported as change in age-normed standard scores (a change of 15 standard score points would represent a change of 1 standard deviation in the general population).The Basic Reading score is a normed composite of the WJ-III subtests Letter-Word Identification and Word Attack, representing word-level reading skill.
Time Frame: 0 and 15 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NF-Tutoring Program 1 | NF-Tutoring Program 2 | Typically Developing Readers | IRD- Tutoring Program 1 | IRD-Tutoring Program 2 | Waitlist Control
Number analyzed (Participants) | 8 | 9 | 26 | 14 | 18 | 14
units on a scale | 13.50 (13.61) | -1.11 (6.94) | -.115 (5.13) | 5.86 (9.31) | 3.06 (9.93) | .143 (7.97)

2. Secondary Outcome: Neuroimaging Data
Description: Neuroimaging data consists of functional MRI and structural MRI measures.
Time Frame: Collected before and after intervention
Reporting Status: Not Posted, anticipated posting 2027-01

ADVERSE EVENTS:
Groups:
- IRD-Tutoring Program 1: These are children with reading disabilities (without NF - ideopathic reading disabilities; IRD) who received Tutoring Program I Tutoring Program I: Tutoring Program I is a structured multi-sensory program that is designed to gradually present the range of sounds and letters with focus on accuracy of phonological concepts and application of those concepts in phrases and sentences. The instruction uses a sequenced defined lesson plan with accuracy and automaticity criteria for skill progression. A range of manipulative and kinesthetic activities is outlined to maintain learner engagement in the intensive intervention design.
Arm/Group | NF-Tutoring Program 1 | NF-Tutoring Program 2 | Typically Developing Readers | IRD-Tutoring Program 1 | IRD-Tutoring Program 2 | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/26 | 0/14 | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/26 | 0/14 | 0/18 | 0/14

LIMITATIONS AND CAVEATS:
Small sample size; Different group sizes; Random assignment to treatment group (along with small sample size) produced some asymmetry of pretest score by treatment group, such that the NF-Tutoring Program 2 started with a higher group mean score.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No